CLINICAL TRIAL: NCT02570906
Title: A Performance Assessment of a Remote Patient Monitoring Device in Measuring Heart Rate, Respiration Rate, Posture, and Activity Level
Brief Title: Performance Assessment of a Remote Patient Monitoring Device
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPO0517; NCT02606968 (obsolete NCT alias)
Record Dates: First submitted 2015-09-01; First posted 2015-10-07 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Physiologic Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Zephyr BioPatch — Remote patient monitoring devices: BioPatch™ (ZephyrLIFE Hospital System™)

SUMMARY:
This study will evaluate the performance of the Zephyr BioPatch in measuring heart rate, respiration rate, posture, and activity level compared to reference devices in healthy adult subjects during a variety of situations including hospital room movements, talking, and a short bout of exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent by subject or legally authorized representative (LAR)
2. Male or female of any race
3. 18-50 years of age, inclusive
4. Willingness to have study devices attached during study participation
5. Willingness to participate in all aspects of the study
6. Ability to walk without human assistance or walking aides (e.g. cane or walker), in the opinion of the investigator

Exclusion Criteria:

1. Subject is unable to provide informed consent
2. Under 18 years of age or over 50 years of age
3. Implanted pacemaker or defibrillator
4. Diagnosis of atrial fibrillation as reported by the subject
5. Current hospital admission
6. History of hospital admission or a surgical procedure in the 60 days prior to study enrollment
7. Any contraindications to protocol specific repositioning techniques (e.g. turning on right side or left side or lying in supine position)
8. Female subject is pregnant and/or lactating as reported by the subject
9. Subject is considered as being morbidly obese (defined as BMI >39.5)
10. Subject is on any medications, in the opinion of the investigator, that would impair heart response during the short bout of exercise
11. A serious concurrent medical or other condition, in the opinion of the investigator, that would impair protocol compliance or safety of the subject

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers, Adults 18 to 50 years old
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Heart rate accuracy | On the day of enrollment to completion of one-time study visit
  No follow-up visits will occur
Heart rate precision | On the day of enrollment to completion of one-time study visit
  No follow-up visits will occur
Respiratory rate accuracy | On the day of enrollment to completion of one-time study visit
  No follow-up visits will occur
Respiratory rate precision | On the day of enrollment to completion of one-time study visit
  No follow-up visits will occur
Activity | On the day of enrollment to completion of one-time study visit
  Activity will be classified as lying, upright, walking, or running.
Body orientation (position) | On the day of enrollment to completion of one-time study visit
  Body orientation (position) if lying horizontally will be classified as facing right, facing left, facing down (prone), or facing up (supine).

CONTACTS AND LOCATIONS:
Overall Officials: William Whang, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States